CLINICAL TRIAL: NCT02885350
Title: Spinal or Epidural Fentanyl or Sufentanil for Labour Pain in Early Phase of the Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Ahonen, MD, Ph.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: §12/19.6.2016/HUS/400/2016; 2016-000486-23 (EudraCT Number)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Results first posted 2021-05-19 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Spinal fentanyl (Active Comparator): 20 micrograms of intrathecally administered fentanyl in single dose. Total volume of intrathecal injection 2 ml.
  Interventions: Drug: Spinal analgesia for labour pain
- Epidural fentanyl (Experimental): 100 micrograms of epidurally administered fentanyl in a single dose. Total volume of epidural injection 7 ml.
  Interventions: Drug: Epidural analgesia for labour pain
- Spinal sufentanil (Active Comparator): 5 micrograms of intrathecally administered sufentanil in a single dose. Total volume of intrathecal injection 2 ml.
  Interventions: Drug: Spinal analgesia for labour pain
- Epidural sufentanil (Experimental): 20 micrograms of epidurally administered sufentanil in a single dose. Total volume of epidural injection 7 ml.
  Interventions: Drug: Epidural analgesia for labour pain

INTERVENTIONS:
Drug: Spinal analgesia for labour pain — Intrathecal dose of either fentanyl or sufentanil delivered by combined spinal-epidural technique
  Arms: Spinal fentanyl; Spinal sufentanil
Drug: Epidural analgesia for labour pain — Epidural dose of either fentanyl or sufentanil delivered through an epidural catheter.
  Other Names: labor epidural; labour epidural
  Arms: Epidural fentanyl; Epidural sufentanil

SUMMARY:
In this study the analgesic effect of two different opioids (fentanyl and sufentanil) will be compared when given either intrathecally or epidurally in primiparous parturients during early phase of the labour.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous parturients
* In early phase of labour (cervical dilatation at or under 5 cm)
* No prior opioids by any route of administration within past 120 min
* Pain at or over 80 mm on 0-100 mm visual analog scale during contraction

Exclusion Criteria:

* Allergy for any of the medications used
* Contraindications for epidural/spinal analgesia
* BMI at the time of delivery under 20 or over 35 kg/m2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antti J Vaananen, M.D., Ph.D., Principal Investigator — Helsinki University Central Hospital (Katiloopiston sairaala)
Locations (1):
- Maternity Hospital, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vaananen A, Kuukasjarvi M, Tekay A, Ahonen J. Spinal and epidural sufentanil and fentanyl in early labour. Acta Anaesthesiol Scand. 2019 Nov;63(10):1413-1418. doi: 10.1111/aas.13450. Epub 2019 Jul 23. PMID 31286476

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Fentanyl | Epidural Fentanyl | Spinal Sufentanil | Epidural Sufentanil
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Parturients in active labour
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Fentanyl | Epidural Fentanyl | Spinal Sufentanil | Epidural Sufentanil | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 20 | 80
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 20 | 20 | 20 | 20 | 80
Pain visual analog scale at 0-100 mm [Mean (Standard Deviation); unit: mm] — A 100 mm visual analog scale (VAS) is used, where 0 mm presents no pain at all and 100 mm presents the worst possible pain.
  mm | 84 (12) | 87 (9) | 86 (8) | 87 (11) | 86 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change of Maximum Pain During Contraction at 20 Minutes After the Study Drug Delivery
Description: All parturients are to have a pain visual analog scale (VAS - on a 0-100 mm scale) at 80mm or higher before the initial study drug delivery. On this scale 0 mm presents a totally pain free condition while 100 mm presents the worst imaginable pain. The change of maximum pain in millimeters on the VAS scale during the 20 minutes following the study drug delivery will be recorded.
Time Frame: 20 minutes
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Spinal Fentanyl | Epidural Fentanyl | Spinal Sufentanil | Epidural Sufentanil
Number analyzed (Participants) | 20 | 20 | 20 | 20
mm | 60 [46 to 74] | 36 [24 to 47] | 67 [54 to 81] | 42 [30 to 55]

2. Secondary Outcome: The Duration of Labour Analgesia After the Single Dose of Epidural or Intrathecal Opioid
Description: The time from the study drug dose to the administration of next epidural bolus, up to five hours. After the study drug dose all parturients wil have epidural catheters in place for subsequent analgesia.
Time Frame: The data below report an average duration of time that is typically less than three hours
Measure: Mean (95% Confidence Interval); unit: min
Arm/Group | Spinal Fentanyl | Epidural Fentanyl | Spinal Sufentanil | Epidural Sufentanil
Number analyzed (Participants) | 20 | 20 | 20 | 20
min | 177 [121 to 234] | 112 [80 to 143] | 151 [111 to 192] | 130 [93 to 168]

ADVERSE EVENTS:
Time Frame: 30 minutes
Description: The parturient is monitored for 30 minutes after the intervention
Arm/Group | Spinal Fentanyl | Epidural Fentanyl | Spinal Sufentanil | Epidural Sufentanil
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 18/20 | 8/20 | 12/20 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Fentanyl (N=20) | Epidural Fentanyl (N=20) | Spinal Sufentanil (N=20) | Epidural Sufentanil (N=20)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (18) | 8 (8) | 12 (12) | 8 (8) — Opioid induced pruritus

LIMITATIONS AND CAVEATS:
No known limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02885350/Prot_SAP_001.pdf